CLINICAL TRIAL: NCT03395782
Title: Factors Determining End-tidal O2 Concentration in During Pre-oxygenation
Brief Title: Factors Determining Oxygen Wash in During Pre-oxygenation
Status: Completed | Type: Observational
Sponsor: Region Västmanland (Other)
Responsible Party: Principal Investigator, Lennart Edmark, Principal Investigator, Region Västmanland
Other Study IDs: 20170517-184
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Airway Complication of Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Arteriell blood-gases.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Age group 40-49: 30 patients will be stratified to this age group.
- Age group 50-59: 30 patients will be stratified to this age group.
- Age group 60-69: 30 patients will be stratified to this age group.
- Age group 70-79: 30 patients will be stratified to this age group.

SUMMARY:
Earlier studies has shown a correlation between older age and longer time for the rise in the end-tidal O2 concentration during pre-oxygenation. In this study the investigators aim to analyse this correlation more closely and investigate if the arterial partial pressure of oxygen (PaO2) as measured before the start of pre-oxygenation, with the patient breathing air, is a better predictor than age for estimating the time necessary for achieving the goal of pre-oxygenation.

DETAILED DESCRIPTION:
Before induction of general anaesthesia pre-oxygenation is a recommended procedure to enhance the time available for solving a problem with the airway or intubation during induction. This can be accomplished by letting the patient breath normal tidal volumes with 100% oxygen for 3 to 5 minutes during pre-oxygenation. If there is airway closure during tidal volume breathing, pre-oxygenation needs longer time to achieve a maximum effect. Airway closure increases with advanced age and a few earlier studies has also shown a correlation between older age and longer time for the rise in the end-tidal O2 concentration during pre-oxygenation.

Pre-oxygenation is a strongly recommended safety procedure before starting anaesthesia but has at least one major side affect: it is the main reason for the development of atelectasis in the lungs during anaesthesia. Atelectasis impairs oxygenation during anaesthesia and probably increase the risk for postoperative pulmonary complications.

Postoperative complications are more common with advanced age and it is important to understand the mechanisms and risk factors involved.

In this study, the investigators hypothesise that the PaO2 as measured before the start of pre-oxygenation, with the patient breathing air, is a better predictor than age for estimating the time necessary for achieving the goal of pre-oxygenation. If this assumption is correct it might have implication for how pre-oxygenation should be adjusted with advancing age.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for general anaesthesia in American Society of Anesthesiology (ASA) physical status classification grade I-III.
* Body mass index over 18.5 and less than 30 kg/m2
* Peripheral oxygen saturation 92% or more on air.

Exclusion Criteria:

* ASA IV.
* Patients with active smoking and former smokers with a history of smoking more than 6 pack-years.
* Chronic obstructive lung disease.
* Bloodgas with PaO2 ≤ 8 kilopascal (kPa) or PaCO2 ≥ 6.5 kPa.
* Continuous positive airway pressure treatment at night.
* Heart failure or angina pectoris.
* Hemoglobin value less than 100 g/L.
* Pregnancy.
* Any neuromuscular or neurologic illness reducing ventilatory capacity.
* Any endocrine disease influencing basic metabolic demand.
* Not possible to achieve a tight mask seal.
* Patient unable to follow instructions.

Ages: 40 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery in general anaesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
PaO2 breathing air before start of pre-oxygenation and the rise in end-tidal O2 during pre-oxygenation. | 5 minutes.
  An arterial bloodgas with the patient in the supine position breathing air will be analysed with regards to PaO2 and correlated to the rise in end-tidal O2 concentration during pre-oxygenation.

SECONDARY OUTCOMES:
Age and the rise in end-tidal O2 during pre-oxygenation. | 5 minutes.
  Age will be correlated to the rise in end-tidal O2 during pre-oxygenation.

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Edmark, Ph.D., Principal Investigator — Region Västmanland
Locations (1):
- Köping County Hospital, Köping, Västmanland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kang H, Park HJ, Baek SK, Choi J, Park SJ. Effects of preoxygenation with the three minutes tidal volume breathing technique in the elderly. Korean J Anesthesiol. 2010 Apr;58(4):369-73. doi: 10.4097/kjae.2010.58.4.369. Epub 2010 Apr 28. PMID 20508794
- [Result] Sum Ping SJ, Makary LF, Van Hal MD. Factors influencing oxygen store during denitrogenation in the healthy patient. J Clin Anesth. 2009 May;21(3):183-9. doi: 10.1016/j.jclinane.2008.07.004. PMID 19464611
- [Result] Milic-Emili J, Torchio R, D'Angelo E. Closing volume: a reappraisal (1967-2007). Eur J Appl Physiol. 2007 Apr;99(6):567-83. doi: 10.1007/s00421-006-0389-0. Epub 2007 Jan 20. PMID 17237952
- [Result] Gambee AM, Hertzka RE, Fisher DM. Preoxygenation techniques: comparison of three minutes and four breaths. Anesth Analg. 1987 May;66(5):468-70. No abstract available. PMID 3578856
- [Derived] Larsson A, Ostberg E, Edmark L. Arterial partial pressure of oxygen as a marker of airway closure does not correlate with the efficacy of pre-oxygenation: A prospective cohort study. Eur J Anaesthesiol. 2023 Sep 1;40(9):699-706. doi: 10.1097/EJA.0000000000001869. Epub 2023 Jun 30. PMID 37395501